CLINICAL TRIAL: NCT06504888
Title: Influence of Penicillin-allergy on Sinus Lift Procedures: a Retrospective Study
Brief Title: Do Penicillin-allergic Patients Presents a High Risk of Sinus Lift Failure
Status: Recruiting | Type: Observational
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor
Other Study IDs: CIR-ELC-2021-06
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Maxillary Sinus Disease
Keywords: Penicillin allergy; Dental implant; Sinus lift failure
MeSH Terms: interventions — Penicillins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients allergic to penicillin: Patients who cannot take any type of penicillin, who have undergone a lateral sinus lift with simultaneous or delayed dental implant.
- Patients who are not allergic to penicillin: Patients who can take some type of penicillin, who have had a lateral sinus lift with simultaneous or delayed dental implant.
  Interventions: Drug: Penicillin

INTERVENTIONS:
Drug: Penicillin — Compare whether there is a higher incidence of sinus elevation in patients allergic to penicillin compared to non-allergic patients, evaluating clinical histories.
  Other Names: Sinus lift procedure
  Groups: Patients who are not allergic to penicillin

SUMMARY:
This retrospective study aims to evaluate clinical histories to determine if there is a relationship between patients allergic to penicillin and sinus lift failure and the possible post-operative complications that may arise.

DETAILED DESCRIPTION:
Introduction: It is known that patients allergic to penicillin have a tendency to have greater failure of dental implants. It is believed that when prescribing non-penicillin antibiotics, such as clindamycin, the bacterial spectrum is not as wide as penicillin, and it is commonly associated with more drug-resistant microorganisms, such as Cloastridium difficile.

However, this statement, which is well studied in implants, has not been studied as much in sinus lift as a surgical technique.

Objectives

* Primary objectives: For that reason, the primary objective of this study is to evaluate retrospectively, if penicillin allergic patients presents higher risk of failure in lateral sinus lift procedure compared to none-allergic penicillin patients.
* Secondary objectives: Evaluate the differences, in terms of implant failure and intraoperative and post-operative sinus lift complications, between patients allergic to penicillin and those who are not allergic.

Materials and Methods: This retrospective study analyzed patients undergoing lateral sinus lift and rehabilitated with dental implants between the years 2004 and 2024 at the dental clinic of Universitat Internacional de Catalunya, Barcelona (UIC). This study will include adult patients in whom a lateral sinus lift with simultaneous or delayed implants was performed at the university. The clinical history should determine whether or not you are allergic to penicillin, the possible pre- and post-operative complications of the surgical intervention and the evaluation regarding the sinus lift surgery (whether it fails or not) and the subsequent placement of the implant.

ELIGIBILITY:
Inclusion Criteria: men and women over 18 years of age, patients undergoing at least one sinus lift procedure with simultaneous or deferred placement of implants; and patients' containing the following data: (1) Penicillin allergy: presence or absence; (2) Prescribed antibiotic guidelines; (3) Intraoperative complications: no complications, Schneider membrane's perforation; (4) Postoperative complications: No complications, fistula, infection, unspecific failure, hemorrhage, healing by second intention; (5) Results of sinus lift procedure: failure or not; (6) Results of implant placement: failure or not.

Exclusion Criteria: (1) Medical history that was not fully complied with; (2) Patients who did not attend follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing lateral sinus lift and rehabilitated with dental implants
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2004-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maxillary sinus lift procedure failure | 2 years
  "Inability to place the implant after sinus lift"

SECONDARY OUTCOMES:
Implant survival rate | 1 year after implant placement
  "The implant is still in mouth"
Post-operative complications | 1-2 weeks after surgery
  Fistula, infection, unspecific failure, hemorrhage or healing by second intention
Intra-operative complications | In the surgery
  Schneider membrane's perforation: 1-2mm, 2-5mm, 5-10mm or >10mm

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain